CLINICAL TRIAL: NCT03579745
Title: Evaluation of Profile Changes and Torque Control in Dental Bimaxillary Proclination Cases Using Lingual Lever Arm Mechanics vs Conventional Lingual Orthodontic Mechanics A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Kandil, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AKandil
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Bimaxillary Proclination
Keywords: lingual orthodontics; Lever arm; En masse retraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional lingual mechanics (Active Comparator)
  Interventions: Procedure: Lingual orthodontics
- Lever arm lingual mechanics (Experimental)
  Interventions: Procedure: Lingual orthodontics

INTERVENTIONS:
Procedure: Lingual orthodontics — A coil spring will be attached from the lever arm to the first molar tube
  Other Names: Conventional lingual mechanics

SUMMARY:
This study evaluates the profile changes and torque control using lingual lever arm vs conventional lingual mechanics. Half of the patients will receive lever arms and the other half will receive conventional lingual orthodontics.

DETAILED DESCRIPTION:
Conventional lingual orthodontic biomechanics leads to torque loss during en masse retraction of the anterior segment in the bimaxillary proclination cases treated by first premolar extraction. Torque loss affects the final outcome of the treatment negatively.

Adding a lever arm to the lingual wire will transmit the point of force application at or apical to the center of rotation which will reduce or eliminate toqrue loss during anterior segment retraction.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patients with age range 18-30 yrs old.
* Class I bimaxillary dentoalveolar proclination.
* Full permanent dentition.
* Good oral hygiene.
* Maximum anchorage is required.
* Healthy bone around the first molars is needed.

Exclusion Criteria:

.Systemic disease.

* Severe crowding.
* Extracted or missing upper permanent tooth/teeth (except for third molars).
* Signs, symptoms or previous history of temporomandibular disorders (TMD).
* Previous orthodontic treatment.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Nasolabial angle | 12 months
  Soft tissue lateral cephalometric radiograph measurement
Profile convexity reduction | 12 months
  N'-sn -Pog' soft tissue angle

SECONDARY OUTCOMES:
Torque control | 12 months
  U1 - Palatal plane angle

CONTACTS AND LOCATIONS:
Overall Officials: Amr Abuelezz, Professor, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: No